CLINICAL TRIAL: NCT06613308
Title: Association Between Respiratory Tract and Gut Microbiome and the Efficacy and Safety of PD-1/PD-L1 Blockade in Resectable Non-small-cell Lung Cancer: a Single-center Cohort Study
Brief Title: Association Between Microbiome and the Efficacy and Safety of PD-1/PD-L1 Blockade in Resectable NSCLC
Status: Not yet recruiting | Type: Observational
Sponsor: Capital Medical University (Other)
Collaborators: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Bin Cao, M.D., China-Japan Friendship Hospital
Other Study IDs: 2022-YJXBF-03-01
Record Dates: First submitted 2024-09-15; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-08

CONDITIONS: Lung Cancer (NSCLC)
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Drug Therapy; Neoadjuvant Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Microbiome in faeces, sputum, swabs, BALF, surgically resected lung lesions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Arm1(Neoadjuvant immunotherapy combined with chemotherapy)
  Interventions: Drug: Neoadjuvant immunotherapy combined with chemotherapy
- Arm2(Neoadjuvant chemotherapy)
  Interventions: Drug: Neoadjuvant chemotherapy

INTERVENTIONS:
Drug: Neoadjuvant immunotherapy combined with chemotherapy — The treatment regimen consisted of a PD-1/PD-L1 monoclonal antibody in combination with a platinum-containing two-agent standard chemotherapy regimen administered every three weeks. Following two to four cycles of therapy, patients who demonstrated no evidence of disease progression were eligible for surgical resection, which was performed within three to four weeks after the conclusion of the last neoadjuvant therapy. Consolidation with a PD-1/PD-L1 monoclonal antibody was initiated within three to eight weeks after surgery and continued every three weeks. The efficacy of the treatment was evaluated according to the irRECIST criteria. Chemotherapy regimens were selected based on tumour histology and investigator judgement. In the event of poor tolerability, patients may switch between cisplatin or carboplatin treatments.
  Groups: Arm1(Neoadjuvant immunotherapy combined with chemotherapy)
Drug: Neoadjuvant chemotherapy — A platinum-containing two-agent standard chemotherapy regimen was administered every three weeks. Following a two-to-four-cycle therapy, if the patients were evaluated without progressive disease, patients undergo surgical resection within three to four weeks of the final neoadjuvant treatment. Postoperative adjuvant chemotherapy is then conducted in accordance with the recommended regimen outlined in the 2022 edition of the CSCO Guidelines for the Diagnosis and Treatment of Non-Small Cell Lung Cancer. The efficacy of the treatment was evaluated in accordance with the RECIST 1.1 criteria.
  The chemotherapy regimens were selected based on the tumor histology and the judgement of the investigators, in accordance with the standard clinical practice. In the event of poor tolerability, patients may switch between cisplatin or carboplatin treatments.
  Groups: Arm2(Neoadjuvant chemotherapy)

SUMMARY:
This study will investigate the relationship between respiratory and gut microbiome and PD-1/PD-L1 immune checkpoint inhibitor efficacy and immune-related adverse events (irAE) in patients with non-small cell lung cancer (Stage IIA-IIIB）

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old;
* first-diagnosed, driver gene-negative non-small cell lung cancer patients with histopathological confirmed diagnosis (Stage IIA-IIIB);
* at least 1 measurable lesion as defined by RECIST version 1.1; an Eastern Cooperative Oncology Group (ECOG) physical status score of 0-1;
* no prior systemic therapy or radiotherapy;
* the patients are eligible for indications for surgical resection and amenable to - neoadjuvant immunotherapy or chemotherapy after multidisciplinary evaluation;
* signing the written consent before enrollment in the study;
* participants need to have adequate pulmonary ventilation and diffusion function to allow surgical resection by pre-enrolment pulmonary function testing;

Exclusion Criteria:

* refusal of participation or inability to give a clear consent;
* requiring treatment with systemic glucocorticoids and other - immunosuppressive agents;
* use of antibiotics within the previous 3 months or the presence of an infectious disease requiring antibiotic therapy;
* probiotics within 3 months prior to enrolment;
* presence of obstructive pneumonia, cancerous cavities, active tuberculosis;
* the presence of bronchiectasis, combined lung infections, pulmonary fibrosis, uncontrolled diabetes mellitus;
* the presence of primary tumors elsewhere;
* receiving chemotherapy or any other cancer treatment prior to enrolment;
* participants with brain metastases confirmed by brain MRI with contrast prior to enrolment;
* active or pre-existing autoimmune disease;
* the presence of uncontrolled comorbidities, including heart failure, uncontrolled hypertension, unstable angina, interstitial lung disease;
* positive test for hepatitis B surface antigen or hepatitis C ribonucleic acid requiring treatment;
* known positive history or positive test results for human immunodeficiency virus or acquired immunodeficiency syndrome (AIDS);
* history of allergy to study drug components;
* women who are pregnant or breastfeeding;
* previous treatment with anti-PD-1, anti-PD-L1, anti-PDL-2, or anti-CTLA-4 antibodies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The neoadjuvant cohort of patients with non-small cell lung cancer (NSCLC) (stages IIA to selective stage IIIB; squamous or non-squamous cell) who are receiving a PD-1/PD-L1 monoclonal antibody in conjunction with platinum-containing two-agent standard chemotherapy (Arm 1) or platinum-containing two-agent standard chemotherapy (Arm 2).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-09-25 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Major pathological response (mPR) | Whithin time from enrollment to surgery
  defined as ≤10% residual live tumor tissue in lung cancer samples resected after neoadjuvant therapy as assessed by the central pathology laboratory.

SECONDARY OUTCOMES:
Pathologic complete response (pCR) | Whithin time from enrollment to surgery
  defined as the absence of live tumour cells in lung cancer specimens resected after neoadjuvant therapy and in all sampled local lymph nodes according to central pathology laboratory assessment. Patients who are not evaluable according to the central pathological assessment (including patients with R2 margins) or who do not have a surgical specimen will not be considered to have achieved a pCR (e.g. remission will be recorded as 'not evaluable' or 'missing', as appropriate).
Disease free survival (DFS) | Whithin 1 year after surgery
  defined as the time from surgery to the first recurrence of disease (local or distant) or all-cause death, whichever occurs first. DFS was captured only for events after surgery.
Overall survival (OS) | Whithin 1 year after enrollment
  defined as time from enrolment to all-cause death
Immune-related adverse event (irAE) | Whithin 1 year after enrollment
  defined as all levels of adverse drug reactions in antitumor immunotherapy that are judged to be related to immune mechanisms, excluding non-specific infusion reactions.
Changes in microbiomics in respiratory tract and gut | Whithin 1 year after enrollment
  Defined as microbial composition, diversity, and functional activity measured by 16S RNA sequencing
Radiological response | Whithin time from enrollment to surgery
  Defined as radiographic change assesed by RECIST 1.1.
Changes in single-cell immune repertoire | Whithin time from enrollment to surgery
  Defined as diversity of immune receptors (e.g. TCR and BCR) for T and B cells in lung tissues

CONTACTS AND LOCATIONS:
Overall Officials: science and technology center, Principal Investigator — China-Japan Friendship Hospital